CLINICAL TRIAL: NCT03592472
Title: A Randomized, Phase 3, Double-blind, Placebo-controlled Study of Pazopanib With or Without Abexinostat in Patients With Locally Advanced or Metastatic Renal Cell Carcinoma(RENAVIV)
Brief Title: A Study of Pazopanib With or Without Abexinostat in Patients With Locally Advanced or Metastatic Renal Cell Carcinoma (RENAVIV)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Xynomic Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: XYN-602
Record Dates: First submitted 2018-06-23; First posted 2018-07-19 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Renal Cell Carcinoma
Keywords: Renal Cell Carcinoma; Progression-free survival; Abexinostat; Pazopanib; RECIST; Cancer therapy
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — pazopanib; abexinostat

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This is a double-blind study. The sponsor, investigators, study coordinators, and the patients will be blinded to the study drug (abexinostat/placebo).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pazopanib plus abexinostat (Experimental): Randomized patients will receive a combination of pazopanib plus abexinostat. The patients will receive pazopanib by mouth (p.o.) daily on Days 1 to 28 of each treatment cycle and will receive abexinostat p.o twice daily (BID) on Days 1 to 4, 8 to 11, and 15 to 18 of every 28-day cycle, 2 doses 4 hours apart. Patients will be instructed to take their once- daily oral dose of pazopanib and BID oral dose of abexinostat at the same time each day.
  Interventions: Drug: Pazopanib; Drug: Abexinostat
- Pazopanib plus placebo (Placebo Comparator): Randomized patients will receive a combination of pazopanib plus abexinostat matching placebo. The patients will receive pazopanib by mouth (p.o.) daily on Days 1 to 28 of each treatment cycle and will receive abexinostat matching placebo p.o BID on Days 1 to 4, 8 to 11, and 15 to 18 of every 28-day cycle, 2 doses 4 hours apart. Patients will be instructed to take their once- daily oral dose of pazopanib and BID oral dose of placebo at the same time each day.
  Interventions: Drug: Pazopanib; Other: Placebo

INTERVENTIONS:
Drug: Pazopanib — All patients will receive pazopanib at a starting dose of 800 mg by mouth (p.o.) daily on Days 1 to 28 of each treatment cycle. Patients should be instructed to take their once- daily oral dose of pazopanib at the same time each morning. Each dose of pazopanib should be taken with an 8 oz/240 mL glass of water either 1 hour before or 2 hours after a meal. Patients should be instructed to swallow the tablets whole and not chew them.
  Other Names: Votrient®
Drug: Abexinostat — The starting dose and schedule of abexinostat will be 80 mg p.o. BID on Days 1 to 4, 8 to 11, and 15 to 18 of every 28-day cycle, 2 doses 4 hours apart. Each dose of abexinostat should be taken with an 8 oz/240 mL glass of water at least half an hour before meals or more than 2 hours after a meal and must be 4 hours apart. Patients should be instructed to swallow the tablets whole and not chew them.
  Other Names: PCI-24781
  Arms: Pazopanib plus abexinostat
Other: Placebo — The starting dose and schedule of abexinostat matching placebo will be 80 mg p.o. BID on Days 1 to 4, 8 to 11, and 15 to 18 of every 28-day cycle, 2 doses 4 hours apart. Each dose of placebo should be taken with an 8 oz/240 mL glass of water at least half an hour before meals or more than 2 hours after a meal and must be 4 hours apart. Patients should be instructed to swallow the tablets whole and not chew them.
  Arms: Pazopanib plus placebo

SUMMARY:
This is a randomized, Phase 3, double-blind, placebo-controlled study of pazopanib plus abexinostat versus pazopanib plus placebo in patients with locally advanced unresectable or metastatic renal cell carcinoma (RCC).

DETAILED DESCRIPTION:
In this randomized, Phase 3, double-blind, placebo-controlled study, patients will be randomized 2:1 to receive either a combination of pazopanib plus abexinostat or pazopanib plus placebo. At the time of disease progression, patient treatment assignment will be unblinded, and those patients randomized to the pazopanib plus placebo treatment arm will have the option of crossing over to receive treatment with a combination of pazopanib plus abexinostat. After providing written informed consent, patients will be screened for study eligibility within 28 days before their first dose of study drug. After screening assessments, patients who are eligible for inclusion in the study will be randomized and receive their first dose of study drug on Cycle 1 Day 1 (C1D1), within 7 days of randomization. A treatment cycle is 28 days in length. Patients may continue to receive study drug until any of the following events: the development of IRC-verified radiographic progression as assessed by RECIST version 1.1, clinical disease progression, unacceptable toxicity, another discontinuation criterion is met, withdrawal of consent, or closure of the study by the sponsor. No maximum duration of therapy has been set.

ELIGIBILITY:
Inclusion Criteria:

To be enrolled in the study, patients will be required to meet all of the following criteria:

* Patients aged ≥ 18 years at time of study entry.
* Patients have histologically confirmed RCC with clear cell component.
* Patients have locally advanced and unresectable or metastatic disease.
* Measurable disease as assessed only by the investigator (not verified by IRC) according to RECIST version 1.1.
* Patients must not have had any prior vascular endothelial growth factor (VEGF) tyrosine kinase inhibitor treatment in either (neo)adjuvant or locally advanced/metastatic setting. Up to 1 line of prior cytokine or immune checkpoint inhibitor treatment is allowed in either the (neo)adjuvant or metastatic setting provided screening scans indicate progressive disease (PD) during or following completion of treatment.
* Patients have Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Patients have adequate baseline organ function.
* Patients have adequate baseline hematologic function
* Patient must be at least 2 weeks from last systemic treatment or dose of radiation prior to date of randomization.

Exclusion Criteria:

Patients who meet any of the following criteria at Screening will not be enrolled in the study:

* Has persistent clinically significant toxicities (Grade ≥ 2; per NCI CTCAE version 5 from previous anticancer therapy (excluding alopecia which is permitted and excluding Grades 2 and 3 laboratory abnormalities if they are not associated with symptoms, are not considered clinically significant by the investigator, and can be managed with available medical therapies).
* Has untreated central nervous system (CNS) metastases. Patients with treated CNS metastases are eligible provided imaging demonstrates no new or progressive metastases obtained at least 4 weeks following completion of treatment. CNS imaging during Screening is not required unless clinically indicated.
* Has an additional malignancy requiring treatment within the past 3 years. Patients with the following concomitant neoplastic diagnoses are eligible: non-melanoma skin cancer, carcinoma in situ, and non-muscle invasive urothelial carcinoma.
* Poorly controlled hypertension, defined as systolic blood pressure ≥ 160 or diastolic blood pressure ≥ 100 mmHg. Use of anti-hypertensives and rescreening is permitted.
* A new pulmonary embolism or deep venous thrombosis diagnosed within 3 months prior to randomization.
* Has a QTcF interval > 480 msec.
* New York Heart Association Class III or IV congestive heart failure.
* Use of prohibited medication within 7 days or 5 half-lives, whichever is shorter, prior to first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 413 (Estimated)
Dates: Start 2018-07-17 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From randomization date to date of first documentation of progression OR death (up to approximately 4 years).
  To compare the PFS between treatment arms. PFS is defined as the time (month) interval between date of randomization and date of radiographic disease progression or death for those without prior evidence of progression, as assessed by blinded Independent Review Committee (IRC) according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

SECONDARY OUTCOMES:
PFS by investigator assessment according to RECIST version 1.1. | From randomization date to date of first documentation of progression OR death (up to approximately 4 years).
  To compare the PFS between treatment arms by investigator assessment. PFS is defined as the time (month) interval between date of randomization and date of radiographic disease progression or death for those without prior evidence of progression, as assessed by IRC according to RECIST version 1.1.
Overall survival (OS) | From progression or end of study, every 3 months follow up until death, patient withdrawal from study follow-up, or study closure, whichever occurs first (up to approximately 4 years).
  OS is defined as the interval between date of randomization and date of death. The main objective was to compare the OS between treatment arms by investigator assessment.
Adverse events by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5 | From Day 1 until end of treatment visit (up to approximately 4 years).
  To characterize the safety profile of pazopanib in combination with abexinostat.
Objective response rate (ORR) | Screening, Cycle 3 Day 1 (C3D1), Cycle 5 Day 1 (C5D1), Cycle 7 Day 1 (C7D1), and on Day 1 of every third cycle (each cycle is 28 days in length) thereafter until end-of-treatment visit (up to approximately 4 years).
  ORR is defined as the proportion of patients with objective evidence of CR or PR by RECIST version 1.1. The main objective was to compare the ORR between treatment arms by investigator assessment.
Duration of response (DOR) | Screening, Cycle 3 Day 1 (C3D1), C5D1, C7D1, and on Day 1 of every third cycle (each cycle is 28 days in length) thereafter until end-of-treatment visit (up to approximately 4 years).
  DOR is defined as the time from the first documentation of response (CR or PR) to the first documentation of objective tumor progression or death due to any cause by RECIST version 1.1. The main objective was to compare the DOR between treatment arms by investigator assessment.
ORR by RECIST version 1.1 in cross-over patient population | Screening, Cycle 3 Day 1 (C3D1), C5D1, C7D1, and on Day 1 of every third cycle (each cycle is 28 days in length) thereafter until end-of-treatment visit (up to approximately 4 years).
  To describe the ORR in patients who cross over to receive pazopanib plus abexinostat at the time of disease progression on pazopanib monotherapy by investigator assessment.
DOR by RECIST version 1.1 in cross-over patient population | Screening, Cycle 3 Day 1 (C3D1), C5D1, C7D1, and on Day 1 of every third cycle (each cycle is 28 days in length) thereafter until end-of-treatment visit (up to approximately 4 years).
  To describe the DOR in patients who cross over to receive pazopanib plus abexinostat at the time of disease progression on pazopanib monotherapy by investigator assessment.
Mean change from Baseline in Functional Assessment of Cancer Therapy Kidney System Index (FKSI-19) scores | First day of treatment Cycle1, Cycle 2, Cycle 6 (each cycle is 28 days in length) until end-of-treatment visit (up to approximately 4 years).
  To assess the impact of pazopanib with or without abexinostat on disease-related symptoms and health-related quality of life (QoL) by investigator assessment. QoL will be assessed by measuring change from baseline in FKSI-19. The FKSI-19 assesses disease-related symptoms experienced in the past 7 days. Patients are asked to respond to 12 questions ("I have a lack of energy," "I feel pain," for example) by using a 5-point scale (0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, 4=very much; possible total score of 0 to 48).
Mean change from Baseline in Functional Assessment of Chronic Illness Therapy (FACIT-F) scores | First day of treatment Cycle1, Cycle 2, Cycle 6 (each cycle is 28 days in length) and at end-of-treatment visit (up to approximately 4 years).
  To assess the impact of pazopanib with or without abexinostat on disease-related symptoms and QoL by investigator assessment. QoL will be assessed by measuring change from baseline in FACIT-F. The FACIT-F scale measures QoL experienced in the past seven days. The measurement consisted of 5 domains (physical well-being, social/family well-being, emotional well-being, functional well-being, and additional concerns) assessed on a 5-point scale (0=not at all; 1=a little bit; 2=somewhat; 3=quite a bit; 4=very much).

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Munster, M.D., Study Chair — University of California, San Francisco; Rahul Aggarwal, M.D., Study Chair — University of California, San Francisco
Locations (38):
- United States (14):
  - University Of UA Cancer Center(UACC)/DH-SJHMC, Phoenix, Arizona
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCSF Helen Diller Family Comphrensive Cancer Center - Hemato, San Francisco, California
  - Norton Cancer Institute, Norton Healthcare Pavilion, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - GU Research Network/Urology Cancer Center, Omaha, Nebraska
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Northwell Health/Monter Cancer Center, Lake Success, New York
  - Mainstreet Physicans Care, Rochester, New York
  - Precision Cancer Research/Dayton Physicians Network - Treatment, Kettering, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - St. Luke's Hospital, Easton, Pennsylvania
  - HOPE Cancer Center of East Texas, Tyler, Texas
  - Medical Oncology Associates, PS (dba Summit Cancer Centers), Spokane, Washington
- China (2):
  - Beijing Cancer Hospital, Beijing
  - Zhongshan Hospital Affiliated to Fudan University, Shanghai
- Italy (9):
  - Fondazione del Piemonte per l'Oncologia_Istituto di Candiolo, IRCCS_ Oncologia Medica, Candiolo
  - A.O. Cannizzaro_UOS Oncologia Medica, Catania
  - IRCCS Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST) UO Oncologia Medica, Meldola (FC)
  - Istituto Europeo di Oncologia_Unità Oncologia Medica Urogenitale e Cervico Facciale, Milan
  - Istituto Nazionale dei Tumori-Fondazione Pascale- SC Oncologia Medica, Napoli
  - Azienda Ospedaliero-Universitaria Maggiore della Carità Novara_SC Oncologia Medica, Novara
  - Istituti Clinici Scientifici Maugeri Spa-SB_ UO Oncologia Medica, Pavia
  - Azienda Ospedaliero Universitaria Pisana_ UO Oncologia Medica Universitaria, Pisa
  - Fondazione Policlinico Universitario A. Gemelli, U.O.C. Oncologia Medica, Roma
- Poland (4):
  - Szpital Specjalistyczny w Brzozowie Podkarpacki Osrodek Onkologiczny, Brzozów
  - Szpitale Pomorskie Sp. z o.o. Oddział Onkologii i Radioterapii, Gdynia
  - Szpital Specjalistyczny im. Ludwika Rydygiera w Krakowie Sp. z o.o. Oddział Onkologii Klinicznej z Pododdziałem Dziennym, Krakow
  - Clinical Research Center Sp. z o.o., Medic-R Sp. K., Poznan
- South Korea (5):
  - National Cancer Center - Center For Prostate Cancer, Goyang-si
  - CHA Bundang Medical Center, CHA University, Seongnam-si
  - Severance Hospital, Yonsei University Health System - Medical Oncology, Seoul
  - Asan Medical Center - University of Ulsan College of Medicin, Seoul
  - Samsung Medical Center - Hematology-Oncology, Seoul
- Spain (4):
  - H.G.U. de Elche, Elche
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - H.U. Virgen de la Victoria, Málaga

IPD SHARING:
Plan to Share IPD: No